CLINICAL TRIAL: NCT06617923
Title: A Phase 2 Study of Senaparib in Combination With Temozolomide in ARID1A Mutation Associated Ovarian Cancer
Brief Title: Study of Senaparib in Combination With Temozolomide in ARID1A Mutation Associated Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Impact Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J2467sIRB; IRB00443678 (Other: Johns Hopkins Medicine IRB)
Record Dates: First submitted 2024-09-19; First posted 2024-10-01 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Ovary Cancer; Fallopian Tube Cancer; Primary Peritoneal Cavity Cancer
Keywords: ovarian; endometrioid; clear cell; ARID1A mutation
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — senaparib; Temozolomide

STUDY DESIGN:
Intervention Model Description: two-stage, non-randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Senaparib 80mg Temozolomide 20mg
  Interventions: Drug: Senaparib; Drug: Temozolomide

INTERVENTIONS:
Drug: Senaparib — Participants will receive orally 80mg daily Days 1-28 of a 28 day cycle.
Drug: Temozolomide — Participants will receive orally 20mg daily Days 1-21 of a 28 day cycle.
  Other Names: TMZ

SUMMARY:
This is a phase 2 study to test the effectiveness (anti-tumor activity) of the combination of the study drugs, Senaparib and Temozolomide, in patients with clear cell or endometrioid ovarian cancers that have ARID1A pathologic variants.

DETAILED DESCRIPTION:
This is a single-arm phase 2, two-stage, non-randomized multicenter Phase 2 study designed to evaluate the clinical activity (response frequency) of senaparib and temozolomide (TMZ) in patients with recurrent or persistent clear cell or endometrioid ovarian cancer.

Up to 18 adult female subjects will be enrolled and receive senaparib 80mg orally daily Days 1-28 and TMZ 20mg daily Days 1-21 of a 28 day cycle. Tumor assessments will be performed every 8 weeks for first 3 cycles then every 12 weeks thereafter until progressive disease is confirmed. Treatment will continue until either unacceptable toxicity, progression of disease, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.
* Pathologically (histologically or cytologically) confirmed diagnosis of recurrent or persistent clear cell or endometrioid ovarian, fallopian tube, or primary peritoneal carcinoma. Histologic documentation (via the pathology report) indicating at least 50% endometrioid or clear cell morphology is required.
* Presence of an ARID1A pathologic variant or likely pathogenic variant identified by next generation sequencing (NGS) tests (per criteria below)

  * Pathogenic or likely pathogenic ARID1A variant identified NGS tests performed by the labs listed on https://ecog-acrin.org/nci-match-eay131-designated-labs will be considered confirmed for the purposes of this study.
  * Pathogenic ARID1A mutation identified by other NGS tests will need to be confirmed by the study PI prior to enrollment.
* All patients must have measurable disease, according to RECIST v1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions) as ≥20 mm with conventional techniques or as ≥10 mm with spiral CT scan, MRI, or calipers by clinical exam. To be considered pathologically enlarged and measurable, a lymph node must be ≥15 mm in short axis when assessed by CT scan or MRI (CT scan slice thickness recommended to be no greater than 5 mm). See Section 12 for the evaluation of measurable disease.

  * Patients who have received radiation must have evidence of measurable disease outside of the radiation field or have documented progression after radiation at the time of enrollment.
* Patients must have received at least two prior cytotoxic regimens or have platinum-resistant (defined as having progressed within 6 months of last platinum therapy) or platinum-refractory (having progressed during primary platinum therapy) disease.

  * Participants can have received no more than 3 prior lines of cytotoxic therapy (any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow).
  * Unlimited prior hormonal therapy, targeted therapy (including immunotherapy) or antiangiogenic therapy will be permitted.
* Patients must have completed prior therapy as detailed below:

  * Prior Therapy Time from last prior therapy to study treatment start date Chemotherapy (except nitrosoureas or mitomycin C) ≥ 28 days; Nitrosoureas or mitomycin C ≥ 42 days; Small molecule inhibitors ≥ 28 days; Monoclonal antibodies ≥ 28 days; Immunotherapy ≥ 28 days; Radiotherapy (RT) ≥ 28 days from last local site RT ≥ 28 days from stereotactic radiosurgery; ≥ 12 weeks from craniospinal ≥50% radiation of pelvis or total body irradiation Radiation related side effects must have resolved prior to study enrollment Endocrine therapy ≥ 7 days
* Ability to take oral medications and not have gastrointestinal illnesses that would preclude absorption of senaparib or TMZ as judged by the treating physician.
* Patients assigned female at birth, age ≥18 years. Because no dosing or adverse event data are currently available on the use of senaparib and TMZ in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Patients must have adequate organ and marrow function as defined below:

  * Absolute Neutrophil Count ≥1,000/microliter (mcL);
  * Differential Differential with no clinically significant morphologic abnormalities on complete blood count (CBC) testing.
  * Manual differential is encouraged, if clinically indicated, and in cases where an automated differential is abnormal.
  * Hemoglobin ≥9 g/dL;
  * Platelets ≥100,000/mcL;
  * aspartate transferase (AST) (SGOT) or Alanine Transaminase (ALT) (SGPT) ≤3 × institutional ULN;
  * Total Bilirubin ≤1.5 × institutional ULN; Direct bilirubin ≤ ULN for subjects with total bilirubin > 1.5 x ULN (patients with isolated indirect bilirubin elevations and a history of Gilbert's Syndrome are eligible)
  * Creatinine -OR- Glomerular Filtration Rate ≤ institutional upper limit normal (ULN) -OR- ≥50 mL/min/1.73 m2 for patients with creatinine levels above institutional ULN
* Because of the potential DNA damaging effects in a developing human fetus with the study treatment, participants of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation including for one month after last dose of senaparib or temozolomide. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Theoretically, CYP3A induction with senaparib use may result in the loss of efficacy in hormonal contraceptives, thus a barrier method of contraception must be used in addition to hormonal contraceptives due to the potential drug-drug interaction with senaparib. Note: All females will be considered to be of childbearing potential unless postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing).
* For patients with known history of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated and the suppressive therapy must not be an excluded concurrent medication.
* Patients with a known history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, the patients are eligible if the patient has an undetectable HCV viral load and the HCV therapy is not an excluded concurrent medication.
* Patients with treated brain metastases are eligible if follow-up brain imaging ≥ 12 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial, with permission of the protocol chair.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.

Exclusion Criteria:

* Prior treatment with a poly ADP ribose polymerase (PARP) inhibitor or temozolomide.
* Patients who are currently receiving or have previously received any other investigational agents within 3 weeks prior to entering the study.
* Patients who have not recovered (CTCAE v5 grade ≤1) from adverse events due to agents administered more than 4 weeks earlier, unless those events are deemed to have returned to baseline, are irreversible, or are unlikely to develop into a life-threatening condition at the permission of the Protocol Chair (e.g., alopecia).
* Patients who have any of the following:

  * A prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).
  * Abnormalities known to be associated with MDS (e.g. del 5q, chr 7 abn) and myeloproliferative neoplasms (MPN) (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing.
  * A prior history of T-cell lymphoblastic lymphoma/lymphoblastic leukemia (T-ALL).
* Patients with clinical or radiographic evidence of bowel obstruction.
* Severe, active comorbidity per the treating investigator's clinical discretion.
* Pregnant or lactating patients.
* Patients with known human immunodeficiency virus (HIV) infection are ineligible because the treatments involved in this protocol may be immunosuppressive, increasing the risk of lethal infections in this patient population.
* Patients with known, untreated brain metastases, as progressive neurologic dysfunction may develop that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to senaparib or temozolomide.
* Strong CYP3A4 inhibitors or inducers should not be used within 3 days of Day 1 dosing until the end of study. Moderate CYP3A4 inhibitors or inducers should be used with caution.

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/ clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.

* Uncontrolled intercurrent illness including, but not limited to, the following:

  * ongoing or active infection, including latent tuberculosis infection,
  * clinically significant GI disease (such as active Crohn's disease or ulcerative colitis),
  * recent or significant cardiovascular disease (defined as any major CV event within the previous 6 months including myocardial infarction, unstable angina, cardiac arrhythmia, stroke, Pulmonary Embolism (PE), or New York Heart Association Class III or IV heart failure),
  * history of liver function abnormality requiring investigation, drug induced liver injury, chronic liver disease, excessive alcohol consumption or chronic alcohol-induced disease,
  * psychiatric illness/social situations that would limit compliance with study requirements, or
  * any other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects of senaparib and temozolomide. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated on study. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with clear cell or endometrioid ovarian, fallopian tube, or primary peritoneal cancer.
Enrollment: 18 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3 years
  Clinical activity (response frequency) of Senaparib and Temozolomide. The primary endpoint of clinical activity is the objective response rate (ORR) defined as complete response (CR) + partial response (PR). Tumor response is defined by RECIST v 1.1. If a patient fails to respond (or has stable disease), the patient will be defined as a non-responder in the analysis. ORR will be estimated using binomial distribution together with 95% Clopper-Pearson confidence interval.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 3 years
  Examine the nature and degree of toxicity in patients treated with this regimen.
  Safety and tolerability will be assessed by clinical review of all relevant parameters including adverse events (AEs), serious AEs (SAEs). Frequency and severity (grades based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0 of AEs will be summarized by system organ class, preferred term, and relation to study drug.
Frequency of Grade 3 and 4 Adverse Events | 3 years
  Number of Grade 3 and 4 treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Gaillard, MD PhD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (2):
- United States (2):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania